CLINICAL TRIAL: NCT03911037
Title: Granulocyte Colony Stimulating Factor Therapy In Decompensated Cirrhosis Of Liver: A Double Blinded Single Centre Randomised Controlled Trial
Brief Title: GCSF Therapy in Decompensated Cirrhosis - A Double Blinded RCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Society for the Study of Liver Diseases, Chandigarh ( India ) (Unknown)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCSF in DC
Record Dates: First submitted 2019-04-06; First posted 2019-04-10 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Decompensated Cirrhosis of Liver
Keywords: Regenerative medicine
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Therapy + G CSF Therapy (Active Comparator): Standard medical therapy will include nutritional support, rifaximin, lactulose, bowel wash, albumin, diuretics, multivitamins, antibiotics. fresh frozen plasma and packed red-cell transfusions (as required). G-CSF ( prefilled syringe) at the dosage of 5 μg/Kg subcutaneously every 12 hr will be administered for five consecutive days. Four such cycles at 3 monthly intervals will be administered.
  Interventions: Drug: G-CSF
- Standard Medical Therapy + Placebo (Placebo Comparator): Standard medical therapy will include nutritional support, rifaximin, lactulose, bowel wash, albumin, diuretics, multivitamins, antibiotics. fresh frozen plasma and packed red-cell transfusions (as required).
  Placebo ( prefilled syringe) filled with normal saline subcutaneously every 12 hr will be administered for five consecutive days. Four such cycles at 3 monthly intervals will be administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: G-CSF — G-CSF will be administered as prefilled syringes at a dosage of 5 μg/Kg subcutaneously every 12 hr for five consecutive days. Four such cycles will be administered at three monthly intervals.
  Arms: Standard Medical Therapy + G CSF Therapy
Drug: Placebo — Placebo ( prefilled syringe) filled with normal saline subcutaneously every 12 hr will be administered for five consecutive days. Four such cycles at 3 monthly intervals will be administered.
  Arms: Standard Medical Therapy + Placebo

SUMMARY:
Cirrhosis of liver is a leading cause of morbidity and mortality worldwide. Complications like ascites, spontaneous bacterial peritonitis, variceal bleed, hepatic encephalopathy, hepatorenal syndrome (HRS) and hepatocellular carcinoma (HCC) portend a poor prognosis and further decreases survival in these patients. The major causes of cirrhosis include excessive alcohol consumption, viral hepatitis and non- alcoholic fatty liver disease.

Currently the only definitive treatment option for cirrhosis is liver transplantation which is limited in its applicability due to donor shortage, exorbitant costs and lack of widespread availability. Moreover, it requires lifelong immunosuppression and has considerable long term side effects including chronic renal failure, post-transplant lymphoproliferative disease and cardiovascular complications.

The ability of stem cells to differentiate into multiple cellular lineages makes one speculate that stem cells can be used for tissue repair and regeneration when tissue-resident stem cells become overwhelmed. It has been shown that in response to acute or chronic liver damage, bone marrow derived stem cells can spontaneously populate the liver and differentiate into hepatic cells, thereby contributing to hepatic regeneration. Thus, apart from hepatocytes and intrahepatic stem cells, bone marrow derived stem cells also participate in the liver regeneration process.

Currently, there are two methods to mobilize stem cells from the bone marrow to the liver. One is administration of cytokines like granulocyte-colony stimulating factor (G-CSF) and the other is the isolation of stem cells from the marrow and their injection into the hepatic artery or portal vein after purification. The latter is probably more cumbersome and may be potentially risky due to the underlying coagulation abnormalities in cirrhotic patients. Improved liver histology and survival has been noted in patients with cirrhosis following mobilization of bone marrow stem cells by granulocyte-colony stimulating factor (G-CSF).

Three recent studies have demonstrated G-CSF induced mobilization of bone marrow stem cells (CD34 cells) in peripheral blood and their subsequent increase in liver tissue and improved survival in patients with alcoholic hepatitis and ACLF. However, there is a paucity of data on whether G-CSF improves survival and prognosis in patients with decompensated cirrhosis.

Verma, Singh et al have shown in an open label trial that there was significantly better 12 month transplant free survival in ( GCSF+ Growth hormone + standard medical therapy group ) and ( G CSF + standard medical therapy group ) as compared to standard medical therapy group alone. CD 34+ cells at day 6 of therapy increased as compared to baseline. There was also a significant decrease of clinical scores, improvement in nutrition, better control of ascites, reduction in liver stiffness, lesser episodes of infection as well as improvement in QOL scores in the treatment groups having G CSF as compared to baseline.

In a recent study by Newsome et al, a multicentre, open label randomized phase 2 trial, patients were randomized to standard care, treatment with subcutaneous G CSF or treatment with G CSF for 5 days followed by leukaphersis and IV infusion of CD 133 positive haematopoietic stem cells. They did not find any difference in MELD score over time in all 3 treatment groups. Serious adverse effects were more common in the G CSF groups than in standard treatment group.

In a study by Kedarisetty CK et al. a significantly larger proportion of patients with decompensated cirrhosis given a combination of G-CSF & Darbopoietin α survived for 12 months more than patients given only placebo ( 68% vs. 26.9%; P = 0.001 ). The combination therapy also reduced liver severity scores and sepsis to a greater extent than placebo.

In view of the conflicting results of the above studies and no studies on the use of multiple courses of GCSF in patients with decompensated cirrhosis in a double blind manner, the present study was undertaken to assess the safety and efficacy of G-CSF in patients with decompensated cirrhosis in the form of a double blinded RCT.

ELIGIBILITY:
Inclusion Criteria:

• Decompensated Cirrhosis of liver irrespective of etiology

Exclusion Criteria:

* Acute on chronic liver failure (fulfilling either APASL or CANONIC criteria of ACLF)
* Splenic diameter of more than 18 cm
* Concomitant HCC or other active malignancy
* Upper gastrointestinal bleeding in the previous 7 days
* Portal vein thrombosis
* Severe renal dysfunction as defined by creatnine > 1.5mg/dl
* Severe cardiac dysfunction
* Uncontrolled diabetes (HbA1c ≥ 9) or diabetic retinopathy
* Acute infection or disseminate intravascular coagulation
* Active alcohol abuse in last 3 months
* Known hypersensitivity to G-CSF
* HIV co-infection
* Pregnancy
* Refusal to give informed consent
* Those opting for liver transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-04 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | One year
  Overall Survival at 1 year from the onset of therapy

SECONDARY OUTCOMES:
Hemopoietic stem cell mobilisation | One Year
  Mobilisation of CD 34+ cells in peripheral blood
Clinical improvement in liver functions | One Year
  Occurrence of decompensations namely ascites, hepatic encephalopathy and variceal bleed
Biochemical improvement in liver functions | One Year
  Improvement in model for end-stage liver disease (MELD) score. MELD score includes serum bilirubin, serum creatinine and international normalized ratio (INR). The score ranges from 6 to 40 with higher score indicating more severe liver disease.
Improvement in nutritional status | One Year
  Nutritional status will be assessed by skeletal muscle index (SMI) measurement using CT scan measurements at L3 level
Improvement in quality of life | One year
  Quality of life will be assessed using SF-36V2 Health Survey questionnaire
Depression | One year
  Improvement in Depression as assessed by Patient Health Questionnaire (PHQ-9). The questionnaire score ranges from 1 to 27 with 1 indicating minimal depression and 27 indicating severe depression.
Demoralisation scale | One year
  Change in demoralisation scale will be noted at baseline and at the end of one year. The demoralisation scale is a questionnaire comprising of 24 items each being scored from 0 to 4. The total score ranges from 0 to 96 with higher score indicating more severe demoralisation.
Immunological profile | One year
  Change in the immunological profile of patients. Immunological profile will be assessed using various interleukins (IL) including IL-6, IL-10, TNF-alpha, IL-17, IL-4, IL-13 and IFN-gamma which will be measured in pg/ml at baseline and at the end of one year.
Safety of G-CSF as assessed by its adverse effects | One year
  Safety of G-CSF as assessed by its adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venkitaraman A, De A, Verma N, Kumari S, Leishangthem B, Sharma RR, Kalra N, Grover S, Singh V. Multiple cycles of granulocyte colony-stimulating factor in decompensated cirrhosis: a double-blind RCT. Hepatol Int. 2022 Oct;16(5):1127-1136. doi: 10.1007/s12072-022-10314-x. Epub 2022 Mar 23. PMID 35322373